CLINICAL TRIAL: NCT06207188
Title: Identification and Differentiation of Thyroid Nodules by Acoustic Imaging and Viscoelastic Parameters
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 08-008778; R01CA148994 (NIH); NCI-2023-10842 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 08-008778 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-01-03; First posted 2024-01-16 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Thyroid Gland Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients undergo ultrasound imaging on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study is being done to identify and differentiate thyroid nodules by acoustic imaging and viscoelastic parameters.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identification of thyroid nodules by vibro-acoustography - Determine detection rate.

II. Evaluate the specificity of VA in differentiating malignant and benign of thyroid nodules - Compare the result to that of ultrasound (US).

III. Assess diagnostic value of Shear Wave Ultrasound Vibrometry (SDUV) and Comb Push shear elastography (CUSE) in differentiation of thyroid nodules - correlate SDUV and CUSE results to pathology.

IV. Test and compare the results shear wave imaging with new FDA approved ultrasound device called SuperSonic Imagine Aixplorer.

V. Assess diagnostic value of Shear Wave Ultrasound Vibrometry (SDUV) and Comb Push shear elastography (CUSE) in differentiation of palpable and sonographically detectable cervical lymph nodes or non-thyroidal neck masses.

VI. Assess the diagnostic values of ultrasound quantitative microvessel imaging for differentiation of thyroid nodules and cervical lymph nodes.

VII. Assess the response to alcohol ablation on patients with recurrent thyroid cancer on thyroid bed or new lymph nodes on neck.

OUTLINE: This is an observational study.

Patients undergo ultrasound imaging on study.

ELIGIBILITY:
Inclusion Criteria:

* * Male and female patient volunteers ages 8 and up who are suspicious for thyroid cancer

  * Patients who have palpable and sonographically detectable lymph nodes or nonthyroidal neck masses and are referred to Radiology Department or Endocrinology for fine-needle aspiration biopsy (FNAB)
  * Patients 18 and up who were previously diagnosed with thyroid cancer and treated with thyroidectomy and recently diagnosed as having recurrence nodes on thyroid bed or on their neck

Exclusion Criteria:

* Because thyroid cancer is rare under the age of 8 years, children younger than this age are excluded from the study
* Having FNAB or surgical biopsy on thyroid in less than two weeks for thyroid nodule detection group
* Having FNAB or surgical biopsy on cervical lymph nodes or non- thyroidal masses for this group of patients

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient volunteers ages 8 and up who are suspicious for thyroid cancer or a group of patients who have palpable and sonographically detectable lymph nodes or nonthyroidal neck masses or who were previously diagnosed with thyroid cancer and treated with thyroidectomy and recently diagnosed as having recurrence nodes on thyroid bed or on their neck.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2009-05-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of nodules successfully sited by vibro-acoustography (VA) | Baseline, 3 months post ablation, 6 months post ablation, 12 months post ablation
  Successful nodule localization will be assessed by the review of the VA image relative to the nodule location information from the reference ultrasound (US) image (agree/disagree on location will be determined for each nodule).
Specificity of VA in differentiating malignant and benign of thyroid nodules | Baseline, 3 months post ablation, 6 months post ablation, 12 months post ablation
  Specificity of VA in differentiating malignant and benign of thyroid nodules will be determined by comparing the VA image to the US image.

CONTACTS AND LOCATIONS:
Overall Officials: Azra Alizad, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials